CLINICAL TRIAL: NCT05204602
Title: Safety and Immunogenicity of Third Dose SARS-CoV-2 Vaccine Booster in Patients With Liver Diseases Following Two Doses of Inactivated Vaccines (NMCID-CHESS 2201): a Multicenter Cohort Study
Brief Title: Safety and Immunogenicity of COVID-19 Vaccine Booster in Patients With Liver Diseases
Acronym: NMCIDCHESS2201
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: LanZhou University (Other); Xingtai People's Hospital (Other); The Third Central Hospital of Tianjin (Unknown); The Third People's Hospital of Taiyuan (Other); Lishui Country People's Hospital (Other); Baoding People's Hospital (Unknown); The Affiliated Hospital of Qingdao University (Other); Affiliated Hospital of Nanjing University of Chinese Medicine (Other); The Fifth People's Hospital of Wuxi (Unknown); Jincheng People's Hospital (Other); The Sixth Peoples Hospital of Shenyang (Unknown); Zhenjiang Third Hospital (Unknown); The Third People's Hospital of Linfen City (Unknown); The First Affiliated Hospital of Dalian Medical University (Other); The Fourth People's Hospital of Qinghai Province (Other); The Third People's Hospital of Tibet Autonomous Region (Unknown); The Second Affiliated Hospital of Chongqing Medical University (Other); Peking University Health Science Center (Other); The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Professor, Huashan Hospital
Other Study IDs: CLD-BOOST
Record Dates: First submitted 2022-01-20; First posted 2022-01-24 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Vaccine Reaction; Liver Diseases
Keywords: SARS-CoV-2 vaccine booster; liver diseases; safety; immunogenicity
MeSH Terms: conditions — COVID-19; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies should that patients with chronic liver diseases, cirrhosis, hepatocellular carcinoma and post-liver-trasplant status had lower immunological response to SARS-CoV-2 vaccines than healthy population. Along with the waning of antibody and emerging SARS-CoV-2 variants, a third dose SARS-CoV-2 booster vaccination is now considered as an effective strategy. Previous studies showed good safety and immunogenicity of the SARS-CoV-2 booster vaccination in healthy population. However, the relevant information in patients with liver diseases need further research. This study (NMCID-CHESS 2201) aimed to investigate the safety and immunogenicity of the SARS-CoV-2 booster vaccination in population with chronic liver diseases

ELIGIBILITY:
Inclusion Criteria:

* Previously vaccinated with two doses of SARS-CoV-2 vaccines and planning to get booster vaccination.
* Clinically or pathologically diagnosed with pre-existing liver disease, including: chronic liver diseases, cirrhosis, liver cancer, liver transplant subjects, etc.
* Understanding and willing to comply with the study procedures and provides written informed consent.

Exclusion Criteria:

* Pregnancy or lactation.
* Active or known history of SARS-CoV-2 infection.
* Diseases causing immunosuppressive or immunodeficient status or autoimmune diseases.
* A history of discontinuing anti-HBV agents in recent three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with liver disease who completed the whole-course COVID-19 vaccination and is going to get booster vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02-10 (Estimated); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Rate of neutralizing antibody serological conversion after the booster vaccination | Fourteen to 90 days after the booster vaccine
  Neutralizing antibody serological conversion is defined as a change from seronegative at baseline to seropositive or a four-fold titre increase if the participant was seropositive at baseline.
Number and rate of all solicited and non-solicited adverse events | Up to 28 days after booster vaccine injection
  First 7 days after the booster dose, participants will be required to record and be interviewed for adverse events; from day 8 to day 28 after booster dose, safety data were collected by spontaneous report.

SECONDARY OUTCOMES:
Number and rate of abnormal laboratory testing results after the booster vaccination | Up to 28 days after after booster vaccine injection
  Abnormal laboratory testing results will be record and grade for severity.
Concentration and titre of neutralizing antibody after booster vaccination | Baseline and 14 days, 28 days, 90 days, and 180 days after the booster vaccination
  The results will be generated from competitive binding immuoenzymatic capture chemiluminescence immunoassays

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Baoding people's Hospital, Baoding, Hebei
  - Xingtai People's Hospital, Xingtai, Heibei
  - Nanjing Hospital of Chinese Medicine Affiliated to Nanjing University of Chinese Medicine, Nanjing, Jiangsu
  - The Fifth People's Hospital of Wuxi Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Zhenjiang Third Hospital Affiliated to Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Sixth Peoples Hospital of Shenyang, Shenyang, Liaoning
  - The Fourth People's Hospital of Qinghai Province, Xining, Qinghai
  - the Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Jincheng People's Hospital, Jincheng, Shanxi
  - The Third People's Hospital of Linfen City, Linfen, Shanxi
  - The Third People's Hospital of Taiyuan, Taiyuan, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - The Third Central Hospital of Tianjin, Tianjin, Tianjin Municipality
  - The Third People's Hospital of Tibet Autonomous Region, Lhasa, Tibet
  - Lishui People's Hospital, Lishui, Zhejiang

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Sarin SK, Choudhury A, Lau GK, Zheng MH, Ji D, Abd-Elsalam S, Hwang J, Qi X, Cua IH, Suh JI, Park JG, Putcharoen O, Kaewdech A, Piratvisuth T, Treeprasertsuk S, Park S, Wejnaruemarn S, Payawal DA, Baatarkhuu O, Ahn SH, Yeo CD, Alonzo UR, Chinbayar T, Loho IM, Yokosuka O, Jafri W, Tan S, Soo LI, Tanwandee T, Gani R, Anand L, Esmail ES, Khalaf M, Alam S, Lin CY, Chuang WL, Soin AS, Garg HK, Kalista K, Batsukh B, Purnomo HD, Dara VP, Rathi P, Al Mahtab M, Shukla A, Sharma MK, Omata M; APASL COVID Task Force, APASL COVID Liver Injury Spectrum Study (APCOLIS Study-NCT 04345640). Pre-existing liver disease is associated with poor outcome in patients with SARS CoV2 infection; The APCOLIS Study (APASL COVID-19 Liver Injury Spectrum Study). Hepatol Int. 2020 Sep;14(5):690-700. doi: 10.1007/s12072-020-10072-8. Epub 2020 Jul 4. PMID 32623632
- [Background] Iavarone M, D'Ambrosio R, Lampertico P; CirCoV study group. Reply to: Correspondence on "High rates of 30-day mortality in patients with cirrhosis and COVID-19". J Hepatol. 2020 Dec;73(6):1570-1571. doi: 10.1016/j.jhep.2020.08.001. Epub 2020 Aug 7. No abstract available. PMID 32771429
- [Background] Qi X, Wang J, Li X, Wang Z, Liu Y, Yang H, Li X, Shi J, Xiang H, Liu T, Kawada N, Maruyama H, Jiang Z, Wang F, Takehara T, Rockey DC, Sarin SK; COVID-Cirrhosis-CHESS Group. Clinical course of COVID-19 in patients with pre-existing decompensated cirrhosis: initial report from China. Hepatol Int. 2020 Jul;14(4):478-482. doi: 10.1007/s12072-020-10051-z. Epub 2020 May 22. PMID 32440857
- [Background] Moon AM, Webb GJ, Aloman C, Armstrong MJ, Cargill T, Dhanasekaran R, Genesca J, Gill US, James TW, Jones PD, Marshall A, Mells G, Perumalswami PV, Qi X, Su F, Ufere NN, Barnes E, Barritt AS, Marjot T. High mortality rates for SARS-CoV-2 infection in patients with pre-existing chronic liver disease and cirrhosis: Preliminary results from an international registry. J Hepatol. 2020 Sep;73(3):705-708. doi: 10.1016/j.jhep.2020.05.013. Epub 2020 May 21. No abstract available. PMID 32446714
- [Background] Qi X, Liu Y, Wang J, Fallowfield JA, Wang J, Li X, Shi J, Pan H, Zou S, Zhang H, Chen Z, Li F, Luo Y, Mei M, Liu H, Wang Z, Li J, Yang H, Xiang H, Li X, Liu T, Zheng MH, Liu C, Huang Y, Xu D, Li X, Kang N, He Q, Gu Y, Zhang G, Shao C, Liu D, Zhang L, Li X, Kawada N, Jiang Z, Wang F, Xiong B, Takehara T, Rockey DC; COVID-Cirrhosis-CHESS Group. Clinical course and risk factors for mortality of COVID-19 patients with pre-existing cirrhosis: a multicentre cohort study. Gut. 2021 Feb;70(2):433-436. doi: 10.1136/gutjnl-2020-321666. Epub 2020 May 20. No abstract available. PMID 32434831
- [Background] He Q, Zhang G, Gu Y, Wang J, Tang Q, Jiang Z, Shao C, Zhang H, Chen Z, Ma B, Liu D, Xie G, Xu D, Huang Y, Zhang H, Liang M, Huang H, Wang Y, Liu H, Yang J, Pan H, Zou S, Li F, Wang F, Liu C, Wang W, Xiong B, Li X, Liu L, Yang J, Qi X. Clinical Characteristics of COVID-19 Patients With Pre-existing Hepatitis B Virus Infection: A Multicenter Report. Am J Gastroenterol. 2021 Feb 1;116(2):420-421. doi: 10.14309/ajg.0000000000000924. No abstract available. PMID 32925195
- [Background] Ai J, Wang J, Liu D, Xiang H, Guo Y, Lv J, Zhang Q, Li J, Zhang X, Li Q, Liang J, Guo X, Feng Y, Liu L, Zhang X, Qin W, Wang X, Rao W, Zhang Q, Tian Q, Zhang Y, Xie F, Jiang S, Yan Y, Qiu Y, Wu H, Hou Z, Zhang N, Zhang A, Ji J, Yang J, Huang J, Zhao Z, Gu Y, Bian L, Zhang Z, Zou S, Ji H, Ge G, Du X, Hou A, Zhu Y, Cong Q, Xu J, Zu H, Wang Y, Yan Z, Yan X, BianBa Y, Ci Q, Zhang L, Yang S, Gao X, Zhong L, He S, Liu C, Huang Y, Liu Y, Xu D, Zhu Q, Xu X, Lv M, Zhang W, Qi X. Safety and Immunogenicity of SARS-CoV-2 Vaccines in Patients With Chronic Liver Diseases (CHESS-NMCID 2101): A Multicenter Study. Clin Gastroenterol Hepatol. 2022 Jul;20(7):1516-1524.e2. doi: 10.1016/j.cgh.2021.12.022. Epub 2021 Dec 20. PMID 34942370
- [Background] Rabinowich L, Grupper A, Baruch R, Ben-Yehoyada M, Halperin T, Turner D, Katchman E, Levi S, Houri I, Lubezky N, Shibolet O, Katchman H. Low immunogenicity to SARS-CoV-2 vaccination among liver transplant recipients. J Hepatol. 2021 Aug;75(2):435-438. doi: 10.1016/j.jhep.2021.04.020. Epub 2021 Apr 21. PMID 33892006
- [Background] Wang J, Hou Z, Liu J, Gu Y, Wu Y, Chen Z, Ji J, Diao S, Qiu Y, Zou S, Zhang A, Zhang N, Wang F, Li X, Wang Y, Liu X, Lv C, Chen S, Liu D, Ji X, Liu C, Ren T, Sun J, Zhao Z, Wu F, Li F, Wang R, Yan Y, Zhang S, Ge G, Shao J, Yang S, Liu C, Huang Y, Xu D, Li X, Ai J, He Q, Zheng MH, Zhang L, Xie Q, Rockey DC, Fallowfield JA, Zhang W, Qi X. Safety and immunogenicity of COVID-19 vaccination in patients with non-alcoholic fatty liver disease (CHESS2101): A multicenter study. J Hepatol. 2021 Aug;75(2):439-441. doi: 10.1016/j.jhep.2021.04.026. Epub 2021 Apr 24. PMID 33905793
- [Background] Ai J, Zhang H, Zhang Q, Zhang Y, Lin K, Fu Z, Song J, Zhao Y, Fan M, Wang H, Qiu C, Zhou Y, Zhang W. Recombinant protein subunit vaccine booster following two-dose inactivated vaccines dramatically enhanced anti-RBD responses and neutralizing titers against SARS-CoV-2 and Variants of Concern. Cell Res. 2022 Jan;32(1):103-106. doi: 10.1038/s41422-021-00590-x. Epub 2021 Nov 23. No abstract available. PMID 34815511
- [Background] Cornberg M, Buti M, Eberhardt CS, Grossi PA, Shouval D. EASL position paper on the use of COVID-19 vaccines in patients with chronic liver diseases, hepatobiliary cancer and liver transplant recipients. J Hepatol. 2021 Apr;74(4):944-951. doi: 10.1016/j.jhep.2021.01.032. Epub 2021 Feb 6. PMID 33563499
- [Background] Hillus D, Schwarz T, Tober-Lau P, Vanshylla K, Hastor H, Thibeault C, Jentzsch S, Helbig ET, Lippert LJ, Tscheak P, Schmidt ML, Riege J, Solarek A, von Kalle C, Dang-Heine C, Gruell H, Kopankiewicz P, Suttorp N, Drosten C, Bias H, Seybold J; EICOV/COVIM Study Group; Klein F, Kurth F, Corman VM, Sander LE. Safety, reactogenicity, and immunogenicity of homologous and heterologous prime-boost immunisation with ChAdOx1 nCoV-19 and BNT162b2: a prospective cohort study. Lancet Respir Med. 2021 Nov;9(11):1255-1265. doi: 10.1016/S2213-2600(21)00357-X. Epub 2021 Aug 13. PMID 34391547